CLINICAL TRIAL: NCT04222179
Title: Tzu-chi General Hospital,Hualien County,Taiwan,ROC
Brief Title: One Brand-new Maneuver to Place Nasoenteric Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Jen-Shung Lin, Prıncıpal ınvestıgator, Buddhist Tzu Chi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB106-10-A
Record Dates: First submitted 2020-01-02; First posted 2020-01-09 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Nutrient Intake Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Naso-enteric tube placement (Other): The participants needed nutrition from naso-enteric tube feeding are enrolled into this study. Double-blind was not needed here.
  Interventions: Device: ultrathın esophagogastroduodenoscope

INTERVENTIONS:
Device: ultrathın esophagogastroduodenoscope — Place the naso-enteric tube together with the ultrathin esophagogastroduodenoscope from the same nasal cavity

SUMMARY:
Naso-enteric tube feeding is necessary for certain patients. Many methods are used to place a naso-enteric tube, such as bed-side blind method, fluoroscopy method and guide-wire method. INvestigators aim to introduce a safe, non-expensive and fast method to insert a silicon naso-gastric (NG) tube into the small intestine.

DETAILED DESCRIPTION:
Investigators tied a 1-cm surgical suture at the tip of a 16 French silicon NG tube (120 cm long, cost 5 US dollars). One conventional EGD (diameter 2.8 mm) biopsy forceps was inserted into the lumen as a strengthened stylet. Then investigators inserted a biopsy forceps (diameter 2.0 mm) and protruded a little out of the working channel of an ultrathin EGD scope (Fujinon EG 530 N, diameter 5.9 mm) to grasp the suture. The ultrathin EGD and NG tube were parallelly pushed into a selected nostril after adequate decongestive anesthesia (Epinephrine 0.3% + Lidocaine 5%) into the small intestine as deep as possible to the jejunum.

Being placed to the small intestine as far as possible, the NG tube was released and the ultrathin EGD scope withdrew. When the scope was pulled backwards from the stomach, the shape/layout of a NG-tube could be simultaneously monitored and adjusted. At last, the EGD biopsy forceps (2.8 mm) inside the NG tube was removed. With this method, in real life, a plain film is not necessary to confirm the NG tube position. However, for study purpose, a KUB film was taken to check the NG tube position.

ELIGIBILITY:
Inclusion Criteria:

1. Esophageal obstruction
2. Gastric outlet obstruction
3. Duodenal obstruction
4. Pancreatitis
5. Gastroparesis -

Exclusion Criteria:

* (1)Coagulopathy (2)Deviation of nasal septa (3)Conscious disturbance

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
procedure time | wıthın 20 mınutes
  The procedure times to place the tube are recorded

SECONDARY OUTCOMES:
the tıme of naso-enterıc tube usage | within 90 days
  The tıme of the naso-enteric tube was recorded in day

CONTACTS AND LOCATIONS:
Overall Officials: Jen S Lin, VS, Study Director — Buddhist Tzu Chi General Hospital
Locations (1):
- Tzu-chi Hospital, Hualien City, Hua-lien County, Taiwan

IPD SHARING:
Plan to Share IPD: No